CLINICAL TRIAL: NCT00452543
Title: A Double-Blind, Placebo-Controlled Study of Acamprosate Added to Escitalopram and Behavioral Treatment in Major Depressive Disorder (MDD) With Comorbid Alcohol Abuse/Dependence
Brief Title: Acamprosate Added to Escitalopram and Behavioral Treatment for Comorbid Depression and Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Janet Melissa Witte, Dr., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-P-001592/1
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-06

CONDITIONS: Major Depressive Disorder; Alcohol Abuse; Alcohol Dependence
Keywords: Major depressive disorder; Alcoholism; Alcohol abuse; Alcohol dependence
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism | interventions — Acamprosate; Escitalopram; Practice Management, Medical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram plus acamprosate (Experimental)
  Interventions: Drug: acamprosate; Drug: escitalopram; Behavioral: Medical management
- Escitalopram plus placebo (Placebo Comparator)
  Interventions: Drug: escitalopram; Behavioral: Medical management; Drug: Placebo

INTERVENTIONS:
Drug: acamprosate — Acamprosate 333mg, 2 capsules by mouth (i.e., PO), three times per day (i.e., TID), for 12 weeks.
  Other Names: Campral
  Arms: Escitalopram plus acamprosate
Drug: escitalopram — Escitalopram is given for 12 weeks. Dosing is flexible, starting at 10mg PO once per day (i.e., QD) with the possibility of increasing to 30mg PO QD.
  Other Names: Lexapro
Behavioral: Medical management — Based on the COMBINE study. 1 hour of medical management / behavioral intervention at every study visit (7 times over 12 weeks).
  Other Names: Campral and Lexapro
Drug: Placebo — Placebo, 2 capsules PO TID, for 12 weeks
  Other Names: Campral and Lexapro
  Arms: Escitalopram plus placebo

SUMMARY:
This is a study about treatment for people who suffer from both major depression and alcohol abuse or dependence. The study will examine whether the addition of acamprosate to escitalopram and behavioral interventions will improve outcomes for this population.

DETAILED DESCRIPTION:
Depression and alcohol use disorders contribute to a significant proportion of the burden of disease, in the United States and abroad. Patients who suffer from co-morbid depression and alcohol abuse/dependence have illnesses that are more severe, persistent and costly than people with either depression or an alcohol use disorder alone. The treatment of these patients remains controversial. Several studies have demonstrated that antidepressants can be safe and efficacious in the treatment of depression in people who continue to drink, and it is now considered the standard of care to provide such treatment. Other studies have shown that pharmacotherapy with naltrexone or acamprosate can help reduce drinking in alcoholics without co-morbid depression. A logical extension of these findings would be to study the treatment of depressed alcoholics with dual pharmacotherapy, combining an anti-depressant with a medication aimed at treating the alcohol use disorder. We will conduct a randomized, double-blind, placebo controlled trial of escitalopram plus acamprosate and behavioral treatment vs. escitalopram plus placebo and behavioral treatment in 20 depressed alcoholics. Outcome measures will include depression, alcohol use and global functioning.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV diagnostic criteria for MDD (diagnosis based on Structured Clinical Interview for DSM-IV, Patient Edition; SCID I/P)
2. Written informed consent
3. Men and women aged 18-64 years
4. Current diagnosis of alcohol abuse/dependence as per SCID I/P

Exclusion Criteria:

1. Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment.
2. Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, partner with vasectomy).
3. Known history of serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease.
4. History of seizure disorder, brain injury, any history of known neurological disease (multiple sclerosis, degenerative disease such as ALS, Parkinson disease and any movement disorders, etc.).
5. Clinical or lab evidence of untreated hypothyroidism.
6. History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance use disorders (excluding alcohol and nicotine) active within the last 12 months.
7. Current use of other psychotropic drugs, including current use of benzodiazepines, hypnotics, anticonvulsants. Concomitant use of antihistamine drugs will be allowed. Patients will need to be off all antidepressants for at least two weeks by the time of the baseline visit, and four weeks for fluoxetine, and off benzodiazepines and other psychotropics for at least one week. The decision about whether to taper existing medications should be made by the individual and their primary treater based on clinical care and will not be made for purposes of study enrollment. allowed.
8. Patients who have failed to respond during the course of their current major depressive episode to at least two adequate antidepressant trials. An adequate antidepressant trial is defined as six weeks or more of treatment with escitalopram > 20mg/day or its antidepressant equivalent: (fluoxetine 40mg/day, sertraline > 100 mg/day, paroxetine > 40 mg/day, fluvoxamine > 100 mg/day, citalopram > 40 mg/day, escitalopram > 20 mg/day, venlafaxine > 150 mg/day, and duloxetine > 60 mg/day).
9. Any depression-focused or substance-abuse focused psychotherapy (family or marital counseling would be allowed).
10. Patients who have taken an investigational psychotropic drug within the past year.
11. Need for medical or inpatient detoxification from alcohol. This determination will be made by the screening clinician, based on clinical judgement as in the multicenter STAR*D study (PHRC #2000-P-001955 in accordance with methods used in the multi-center STAR-D study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Witte, MD, Principal Investigator — Massachusetts General Hospital; Nicholas Bolo, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Witte J, Bentley K, Evins AE, Clain AJ, Baer L, Pedrelli P, Fava M, Mischoulon D. A randomized, controlled, pilot study of acamprosate added to escitalopram in adults with major depressive disorder and alcohol use disorder. J Clin Psychopharmacol. 2012 Dec;32(6):787-96. doi: 10.1097/JCP.0b013e3182726764. PMID 23131884

RESULTS

PARTICIPANT FLOW:
Groups:
- Escitalopram Plus Acamprosate: Escitalopram 10-30mg/day plus acamprosate 333mg, 2 tabs tid
- Escitalopram Plus Placebo: Escitalopram 10-30mg/day plus placebo 2 tabs tid that resembles acamprosate
Period: Overall Study
Arm/Group | Escitalopram Plus Acamprosate | Escitalopram Plus Placebo
Started | 12 | 11
Completed | 7 | 5
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram Plus Acamprosate | Escitalopram Plus Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (13) | 43 (14) | 47 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Score on the Hamilton Rating Scale for Depression -- 17 Items (HAM-D-17)
Description: Scores on the HAM-D-17 typically fall into the following ranges: a) Not depressed: 0-7; b) Mildly depressed: 7-15; c) Moderately depressed: 15-25; d) Severely depressed: over 25. A decrease of 50% or more in the Hamilton-D score is considered to be a positive response to treatment, while a score of 7 or less is considered typical of remission. We measure the change in total score from Baseline to Week 12 or week of early termination visit.
Time Frame: From baseline visit to Week 12 (or early discontinuation visit)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Escitalopram Plus Acamprosate | Escitalopram Plus Placebo
Number analyzed (Participants) | 12 | 11
Scores on a scale | -5.6 (8.5) | -7.8 (9.9)

2. Primary Outcome: Total Drinking Days on the Alcohol Timeline Followback (TLFB)
Description: The TLFB assesses recent drinking behavior. On the TLFB, clients retrospectively estimate their daily alcohol consumption in standard drinks over a time period ranging from 7 days to 24 months prior to the interview, and thus the measure provides quantitative estimates of alcohol use. One standard drink on the TLFB was defined as: 12 oz beer (5% alcohol by volume), 5 oz of wine (10-12% abv), 3 oz of fortified wine (16-18% abv), or 1-1.2 oz of hard liquor (86-100 proof; 43-50% abv). We measure the change from Baseline to Week 12 or week of early termination visit.
Time Frame: From Baseline visit to Week 12 (or early discontinuation visit)
Population: Intent to treat sample
Measure: Mean (Standard Deviation); unit: Drinking days
Arm/Group | Escitalopram Plus Acamprosate | Escitalopram Plus Placebo
Number analyzed (Participants) | 12 | 11
Drinking days | 61 (53) [8 to 114] | 61 (86) [-25 to 147]
Statistical Analysis 1: Comparison: Escitalopram Plus Acamprosate vs Escitalopram Plus Placebo; Statistical analyses evaluated the null hypothesis that there would be no difference in the effect of acamprosate vs. placebo on total drinking days.Power analysis was originally based on ITT analysis with 40 subjects, and assumed 30% difference in alcohol consumption (50% vs. 20% reduction in the acamprosate and placebo groups, respectively). With alpha of 0.05, we estimated 74% power to detect a difference between the two groups; Test type: Non-Inferiority or Equivalence — This was a test of non-inferiority between the effects of acamprosate vs. placebo. Power analysis was originally based on ITT analysis with 40 subjects, and assumed 30% difference in alcohol consumption (50% vs. 20% reduction in the acamprosate and placebo groups, respectively). With alpha of 0.05, we estimated 74% power to detect a difference between the two groups. Results would be used to estimate effect size to set the stage for an adequately powered larger study in the future; p < 0.05, Wilcoxon (Mann-Whitney) — Threshold for significance was set a priori at p<0.05

3. Primary Outcome: Total Drinks Consumed Per Week on the TLFB
Description: Total Drinks Consumed per Week on the Time Line Follow Back. We measure the change from Baseline to Week 12 or week of early termination visit.
Time Frame: From Baseline visit to Week 12 (or early discontinuation visit)
Measure: Mean (Standard Deviation); unit: Drinks consumed per week
Arm/Group | Escitalopram Plus Acamprosate | Escitalopram Plus Placebo
Number analyzed (Participants) | 12 | 11
Drinks consumed per week | 15 (13) [2 to 28] | 15 (21) [-6 to 36]
Statistical Analysis 1: Comparison: Escitalopram Plus Acamprosate vs Escitalopram Plus Placebo; Statistical analyses evaluated the null hypothesis that there would be no difference in the effect of acamprosate vs. placebo on total drinks consumed per week.Power analysis was originally based on ITT analysis with 40 subjects, and assumed 30% difference in alcohol consumption (50% vs. 20% reduction in the acamprosate and placebo groups, respectively). With alpha of 0.05, we estimated 74% power to detect a difference between the two groups; Test type: Non-Inferiority or Equivalence — This was a test of non-inferiority between the effects of acamprosate vs. placebo; p < 0.05, Wilcoxon (Mann-Whitney) — This p <0.05 was set a priori

4. Primary Outcome: Total Drinks Consumed Per Drinking Day on the TLFB
Description: Total Drinks Consumed per Drinking Day on the Time Line Follow Back. We measure the change from Baseline to Week 12 or week of early termination visit.
Time Frame: From Baseline visit to Week 12 (or early discontinuation visit)
Measure: Mean (Standard Deviation); unit: Drinks consumed per drinking day
Arm/Group | Escitalopram Plus Acamprosate | Escitalopram Plus Placebo
Number analyzed (Participants) | 12 | 11
Drinks consumed per drinking day | 4 (2) [2 to 6] | 4 (4) [0 to 4]
Statistical Analysis 1: Comparison: Escitalopram Plus Acamprosate vs Escitalopram Plus Placebo; Statistical analyses evaluated the null hypothesis that there would be no difference in the effect of acamprosate vs. placebo on total drinks consumed per drinking day. Power analysis was originally based on ITT analysis with 40 subjects, and assumed 30% difference in alcohol consumption (50% vs. 20% reduction in the acamprosate and placebo groups, respectively). With alpha of 0.05, we estimated 74% power to detect a difference between the two groups; Test type: Non-Inferiority or Equivalence — This was a test of non-inferiority between the effects of acamprosate vs. placebo. Statistical analyses evaluated the null hypothesis that there would be no difference in the effect of acamprosate vs. placebo on total drinks consumed per drinking day. Power analysis is discussed above; p < 0.05, Wilcoxon (Mann-Whitney) — This p<0.05 was set a priori

ADVERSE EVENTS:
Arm/Group | Escitalopram Plus Acamprosate | Escitalopram Plus Placebo
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/11
Other Adverse Events (participants affected / at risk) | 8/12 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram Plus Acamprosate (N=12) | Escitalopram Plus Placebo (N=11)
Hospitalization for alcohol intoxication (Psychiatric disorders) | 1 (1) | 0 (0) — Subject was admitted to a detox unit after found intoxicated and passed out. Subject was discharged 3 days following from the inpatient unit to an outpatient program.
Blockage in the coronary artery (Cardiac disorders) | 1 (1) | 0 (0) — Subject had sudden onset of shortness of breath and chest pain. A blockage was discovered in the coronary artery, requiring that a stent be implanted. The patient was hospitalized for 4 days.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram Plus Acamprosate (N=12) | Escitalopram Plus Placebo (N=11)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Increased gag reflex (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Insomnia (General disorders) | 1 (1) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2)
Urinary respiratory infection (Renal and urinary disorders) | 1 (1) | 0 (0)
GI upset (Gastrointestinal disorders) | 1 (1) | 1 (1)
Soft stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Jaw tightening (General disorders) | 0 (0) | 1 (1)
Dry lips (General disorders) | 0 (0) | 1 (1)
Increased sweating (General disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Tension (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No